CLINICAL TRIAL: NCT01248390
Title: "A Randomized, Controlled, Trial of Interactive Metronome Technology for Remediation of Cognitive Difficulties Following Blast-Related Traumatic Brain Injury"
Brief Title: "Interactive Metronome Technology for Blast-Related Traumatic Brain Injury"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-14853.22
Record Dates: First submitted 2010-11-22; First posted 2010-11-25 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Traumatic Brain Injury; Post-Concussion Syndrome
Keywords: traumatic brain injury; post-concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive Metronome therapy (Experimental): Fifteen one-hour training sessions using Interactive Metronome system, in addition to treatment as usual.
  Interventions: Behavioral: Interactive metronome
- Treatment as Usual (No Intervention): Standard of care symptom management.

INTERVENTIONS:
Behavioral: Interactive metronome — A randomized, controlled investigation into the effects of IM training on a sample of boys with attention deficit disorder showed positive results. Compared to an active control treatment, IM training improved performance on a host of measures, including attention, motor control, language processing, reading, and parental reports of improvements in the regulation of aggressive behavior.16 It should be noted that these cognitive and behavioral functions are common symptom areas in individuals surviving TBI and are likely to be especially affected in cases of blast injury
  Arms: Interactive Metronome therapy

SUMMARY:
The purpose of this research is to see whether adding a new therapy helps people with brain injury focus better and think more clearly. You are being asked to participate in this research study because you have had a brain injury. If you decide to volunteer, you will be in the study for about six months.As a participant, you will be randomly assigned to one of 2 treatment plans. Randomization is a process like flipping a coin and means you will have a chance of being assigned to either of the plans. One group will be given an experimental therapy using a metronome one hour a day, three times a week. A metronome is a device that produces a steady beat. You will need to keep time with the metronome doing several different movements. On each beat, you will be given information both through sound and on a computer screen about whether you were early or late and how far off beat you were. The tempo of the beat will be at 54 beats per minute, so you will need to process the feedback information very quickly to adjust your speed up or down to match the beat. The various movements include things like clapping hands, tapping toes, or alternating between different similar movements. It is hoped that the metronome will help subjects to concentrate better.

DETAILED DESCRIPTION:
The design of this study will be a randomized, controlled trial of Interactive Metronome (IM) treatment compared with treatment as usual in patients with moderate to mild Traumatic Brain Injury (TBI) due to blast. The study will be conducted at the Evans Army Community Hospital at Fort Carson, Colorado . Patients will be randomized to IM training, or to a treatment as usual/wait-list control condition. Patients randomized to receive IM training will complete 15 sessions consisting of approximately 2000 repetitions each. Patients randomized to treatment as usual will be offered the opportunity to receive IM training following the conclusion of the six month study period. Outcome assessment will focus on phase lag and coherence of electroencephalogram (EEG) activity, which are electrophysiological measures of cortical connectivity. Primary outcomes will also include attention and memory functioning, which are measured prior to the start of treatment, one week following the end of treatment and 6 months after treatment ends.

Interactive Metronome (IM) technology is a behavioral feedback operant conditioning system.15 In biofeedback, physiological information is displayed to the patient but with IM information about the patient's behavioral responses is provided to them. Below the investigators provide a detailed description of the behavioral tasks and give some idea as to the program's complexity and operation. IM technology takes advantage of each of the above discussed factors related to neuroplastic processes and integrates them into a single set of tasks that are designed to encourage integrated neuroplastic activity under cognitively demanding circumstances. The computerized feedback is reliable, consistent, timely, and directly correlated with motor output. The feedback is also presented in a rich cognitive and sensory environment that combines instantaneous delivery of simultaneous auditory and visual feedback following the motor response. This information aids the preparation of the upcoming behavioral response. All of this feedback processing and adjustment of behavioral responses must occur in just over a second (1.111 seconds) because the default tempo for IM training is 54 beats per minute. This places a considerable temporal demand upon the attentional, integration, decision making, inhibitory, and motor output operators of the cortex, thereby increasing processing speed and efficiency over the course of training.

ELIGIBILITY:
Inclusion Criteria:

1. Blast-related traumatic brain injury patients at least 3 months post injury with recovery to a Rancho los Amigos level 7 or 8 (alert and oriented).
2. Brain injury documented by at least one of the following:

   i. loss of consciousness, post traumatic amnesia ii. alteration in mental status (dazed/confused), and/or physical evidence of iii.trauma (MRI/CT hemorrhage/contusion)
3. A diagnosis of Postconcussional Disorder or Mild Neurocognitive Disorder Due to a General Medical Condition.
4. Military or Veteran beneficiary
5. Males and females aged 18-55

Exclusion Criteria:

1. Current/prior (last 6 months) unstable medical condition that could affect current brain function (e.g. clear anoxic episode, cardiac arrest, current uncontrolled diabetes)
2. Status post craniectomy prior to cranioplasty (must be 90 days post cranioplasty without surgical complication)
3. Prior History of moderate to severe TBI (not including present injury).
4. Current (last 3 months) active suicidal or homicidal ideation or intent.
5. Current (last month) drug/alcohol abuse or dependence as determined by a score of 5 or higher on the Alcohol Use Disorders Identification Test Consumption (AUDIT-C)
6. Use of benzodiazepine or narcotic medications.
7. Participation in a concurrent drug or treatment trial
8. Must be physically able to complete the treatment tasks (including sensory functions).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-08; Primary Completion 2014-05 (Actual); Study Completion 2016-10-03 (Actual)

PRIMARY OUTCOMES:
Outcome Measure | Six Months Post Treatment
  Determine whether IM training leads to improvements in attention and memory immediately post treatment and at six months in comparison to rehabilitation treatment as usual.

SECONDARY OUTCOMES:
Outcome Measure | Six Months Post Treatment
  Determine whether the addition of Interactive Metronome training leads to better secondary outcomes such as postconcussion symptom status, vocational functioning, and quality of life at 6 months in comparison to treatment as usual.

CONTACTS AND LOCATIONS:
Overall Officials: Renee M Pazdan, MD, Principal Investigator — United States Public Health Service
Locations (1):
- Warrior Recovery Center, Colorado Springs, Colorado, United States

REFERENCES:
- [Result] Nelson LA, Macdonald M, Stall C, Pazdan R. Effects of interactive metronome therapy on cognitive functioning after blast-related brain injury: a randomized controlled pilot trial. Neuropsychology. 2013 Nov;27(6):666-79. doi: 10.1037/a0034117. Epub 2013 Sep 23. PMID 24059443